CLINICAL TRIAL: NCT06748573
Title: A Prospective Study of a Novel Pocket Compression Device to Reduce Pocket Hematoma After Cardiac Implantable Electronic Device Implantation in a High Bleeding Risk Population
Brief Title: Compression Device to Reduce Pocket Hematoma After Cardiac Implantable Electronic Device Implantation in a High Bleeding Risk Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maxime Tijskens (Other)
Collaborators: Merit Medical Systems, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Maxime Tijskens, Principal investigator, Ziekenhuis aan de Stroom
Organization: Ziekenhuis aan de Stroom (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5671
Record Dates: First submitted 2024-12-11; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Pocket Hematoma
Keywords: pocket hematoma; compression device; cardiac implantable electronic device

STUDY DESIGN:
Intervention Model Description: The study is single-center, observational, case-controlled, randomized and prospective trail conducted at the ZAS heart center. Before CIED implantation, patients were randomly assigned in a 1:1 ratio to the study group (SafeGuard FocusTM compression device) or control group (standard care with compressive bandage) using a sealed envelope system.
  Inclusion criteria were all patients above 18 years of age undergoing primo CIED implantation (pacemaker, internal cardiac defibrillator or cardiac resynchronization therapy) with a high bleeding risk (as defined by at least 1 of the following risk factors: age > 75 years, heart failure, kidney failure, antithrombotic use (double antiaggregant therapy or anticoagulation). Exclusion criteria were refusal to participate or mental illness.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (Active Comparator): conventional compression bandage
  Interventions: Device: Conventional bandage
- Study arm (Experimental): Study device (inflatable and see-through)
  Interventions: Device: SafeGuard FocusTM compression bandage

INTERVENTIONS:
Device: SafeGuard FocusTM compression bandage — If randomized to the study group, The study device was applied immediately after pocket closure using following steps:
  * Preparation: cleaning wound and surrounding area.
  * Placement: application of isobetadine gauze and transparent bandage. Study device placement at the level of the pocket.
  * Applying compression: inflation of 60ml of air. If oozing persisted 5ml increments were added (maximum of 120ml) until oozing stopped.
  The study device was gradually deflated by removal of 20ml of air every 2 hours. When oozing occurred 5ml increments were added until oozing stopped. When all air was deflated the study device was left in deflated mode and changed by conventional bandage at discharge.
  Arms: Study arm
Device: Conventional bandage — If randomized to the control group, compressive bandage was applied immediately after pocket closure. The bandage was removed after 6 hours and changed by conventional bandage.
  Arms: Control arm

SUMMARY:
Your doctor has determined that you have an indication for cardiac implantation implantable electronic device (CIED = collective name for pacemaker or defibrillator). Pocket bleeding is a possible complication that occurs in 0.2-16% of cases depending on the definition used. They are an important risk factor for CIED infections (factor 9x). Other possible consequences include prolonged hospitalization risk of stroke due to discontinuation of blood thinners and even death. The main known risk factors for pocket bleeding are advanced age, heart failure, kidney failure, congenital bleeding tendency and the use of blood thinners. Have several measures to reduce the risk of pocket bleeding varying or limited effects shown in the past. Currently the standard treatment consists of applying a conventional pressure bandage at the pocket.However, the lack of targeted compression and lack of standardization has caused this only a limited effect and contributes to patient discomfort. Moreover, let a Conventional pressure dressing does not allow the pocket to be evaluated. The SafeGuard FocusTM compression bandage is a promising new option with several technical features advantages: it can deliver 2x as much pressure as a conventional pressure bandage, the amount pressure can be adjusted according to effect and patient comfort and there is a transparent window so that the surgical wound can always be inspected. This new pressure bandages already used in several countries, but has never been compared until now with a conventional pressure bandage.

DETAILED DESCRIPTION:
Prospective study on the potential benefit of SafeGuard FocusTM compression dressing in preventing pocket bleeding after implantation of a cardiac implantable electrical device in patients with an increased risk of bleeding Introduction You are invited to participate in a research study involving up to 200 patients . The study aims to confirm the effectiveness and safety of the SafeGuard FocusTM compression bandage when compared to the conventional compression bandage. Your participation in the study will last a total of 1 month and will take place during the standard follow-up moments on the day of implantation, the next day and the first check-up after 1 month. So no additional follow-up moments are required. Before you agree to participate in this study, please consider how the study is designed and the potential risks and benefits so that you can make an informed decision. This process is called 'giving consent'.

The implantation procedure is identical in both groups, only the type of pressure bandage applied after the procedure is different.

SafeGuard FocusTM compression bandage:

If randomized to the study group, the SafeGuard FocusTM pressure bandage will be applied immediately after closing the skin according to the following steps:

Preparation: Clean and dry wound and surrounding skin Placement: Apply isobetadine gauze and transparent bandage. Apply SafeGuard FocusTM pressure bandage with balloon placed at CIED pocket.

Starting compression: Fill with 60ml of air. If bleeding persists, add an additional 5 mL each time until bleeding stops (maximum 120 mL).

Deflation Step 1 (after 2 hours): check incision and, if possible, remove 20mL of air Deflation Step 2 (after 4 hours): Check incision and, if possible, remove 20mL of air Deflation Step 3 (after 6 hours): Check incision and, if possible, remove 20mL of air SafeGuard FocusTM is then left on the wound without air until the patient is discharged Then apply a classic plaster

Classic pressure bandage:

If randomized to the control group, a classic pressure bandage will be applied to the pocket for 6 hours. Patients are followed up 2 and 4 hours after the procedure, the day after the procedure and 1 month after the procedure. No additional follow-up moments are required compared to implantations outside the current study.

Follow-up Patients were assessed 2, 4 and 6 hours after procedure, day after procedure and one month after procedure. They were also assessed during any visit in between deemed relevant by the investigator. All patients underwent standard device interrogations, chest radiography and echocardiogram on the day after CIED implantation.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing primo CIED implantation (pacemaker, internal cardiac defibrillator or cardiac resynchronization therapy)
* with a high bleeding risk (as defined by at least 1 of the following risk factors: age > 75 years, heart failure, kidney failure, antithrombotic use (double antiaggregant therapy or anticoagulation

Exclusion Criteria:

* refusal to participate
* mental illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
pocket hematome | 24 hours
  Grade I PH is defined as pocket ecchymosis or small effusion in the absence of swelling or pain. Grade II PH consists of large pocket effusion leading to swelling or pain. Grade III PH is characterized by the need of reoperation and/or hospitalization prolongation and/or interruption of antithrombotic drugs.

SECONDARY OUTCOMES:
pain score | 24 hours
  Visual Analog Scale (VAS) pain score (0-10/10 with 0 = no pain at all; 10= worst possible pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiology, Wilrijk, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No
It can be shared at reasonable request